CLINICAL TRIAL: NCT06697106
Title: Can COX-2 Inhibitor Decrease Stricture Recurrence After Direct Vision Internal Urethrotomy?
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: New Valley University (Other)
Responsible Party: Principal Investigator, Waheed Fawzy Abdelrasol, Lecturer of Urology, Faculty of medicine, New Vally University, New Vally, Egypt, New Valley University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 20241030012
Record Dates: First submitted 2024-11-17; First posted 2024-11-20 (Actual); Last update posted 2024-11-21 (Actual); Status verified 2024-11

CONDITIONS: COX-2 Inhibitor; Meloxicam; Stricture Recurrence; Direct Vision Internal Urethrotomy
MeSH Terms: interventions — Anti-Inflammatory Agents, Non-Steroidal

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Nonsteroidal anti-inflammatory drugs (Experimental): Patients will undergo direct vision internal urethrotomy (DVIU) plus nonsteroidal anti-inflammatory drugs (NSAID) for 3 weeks.
  Interventions: Drug: Nonsteroidal anti-inflammatory drugs
- Control group (Placebo Comparator): Patients will undergo direct vision internal urethrotomy (DVIU) plus a placebo for 3 weeks.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Nonsteroidal anti-inflammatory drugs — Patients will undergo direct vision internal urethrotomy (DVIU) plus nonsteroidal anti-inflammatory drugs (NSAID) for 3 weeks.
  Arms: Nonsteroidal anti-inflammatory drugs
Drug: Placebo — Patients will undergo direct vision internal urethrotomy (DVIU) plus a placebo for 3 weeks.
  Arms: Control group

SUMMARY:
To evaluate the efficacy and safety of nonsteroidal anti-inflammatory drugs (NSAIDs) in preventing urethral stricture recurrence after direct visual internal urethrotomy.

DETAILED DESCRIPTION:
The most common aetiology of urethral strictures is idiopathic, followed by iatrogenic causes, including transurethral resection, urethral catheterization, prostate cancer treatments, and previous hypospadias surgery.

The recurrence rates are higher with previously treated, long and multiple strictures, penile compared with bulbar strictures, and those with perioperative infection.

It has been reported that post-transurethral resection of the prostate (TURP) to receive or not receive a COX-2 inhibitor (rofecoxib 25 mg/day) for 20 days. At 1 year of follow-up, a urethral stricture had been diagnosed in 17 and 0 % of cases without and with COX-2 treatment, respectively

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* American Society of Anesthesiologists (ASA) score ≤3.
* Urethral stricture length ≤ 1.5 cm

Exclusion Criteria:

* Recurrent urethral stricture ≥ 2 times.
* Pelvic fracture urethral distraction defect (PFUDD).

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Males undergoing direct vision internal urethrotomy
Enrollment: 82 (Estimated)
Dates: Start 2024-11-20 (Actual); Primary Completion 2025-04-01 (Estimated); Study Completion 2025-04-01 (Estimated)

PRIMARY OUTCOMES:
Urethral stricture recurrence | 90 days postoperative
  Urethral stricture recurrence is defined as the need for a secondary procedure, including dilation, internal urethrotomy, and urethroplasty, considered as treatment failure.

SECONDARY OUTCOMES:
International Prostate Symptom Score (IPSS) | 90 days postoperative
  The International Prostate Symptom Score (IPSS) will be used to assess lower urinary tract symptoms (LUTS). The IPSS consists of seven questions related to voiding symptoms. A score of 0 to 7 indicates mild symptoms, 8 to 19 indicates moderate symptoms, and 20 to 35 indicates severe symptoms.
Quality of life (QOL) | 90 days postoperative
  Quality of life (QOL) will be used to assess lower urinary tract symptoms (LUTS). Patients will answer using a Likert scale, with four or five response options per item, and scores range from 0 (best QoL) to 13 (worst QoL).
Maximum flow rate | 90 days postoperative
  Maximum flow rate (Q.max) will be used to assess lower urinary tract symptoms (LUTS).
Incidence of complications | 90 days postoperative
  Incidence of complications will be recorded.

CONTACTS AND LOCATIONS:
Locations (1):
- New Valley University, New Valley, New Valley Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Yes
The data will be available upon a reasonable request from the corresponding author after the end of study for one year.
Supporting Information: Study Protocol
Time Frame: After the end of study for one year.
Access Criteria: The data will be available upon a reasonable request from the corresponding author.